CLINICAL TRIAL: NCT03490799
Title: Musculoskeletal Ultrasound Versus Magnetic Resonance Imaging in Assessment of Meniscal Abnormalities.
Brief Title: Muskloskeletal Ultrasound Versus Magnetic Resonance Imaging in Meniscal Abnormalities
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Ali, Principle Investigator, Assiut University
Other Study IDs: MSK US Versus Mri
Record Dates: First submitted 2018-03-31; First posted 2018-04-06 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-03

CONDITIONS: Meniscus Lesion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
clinical examination alone is usually insufficient in assessment of knee meniscus and a more reliable diagnosis can be achieved by using the knee ultrasound , magnetic resonance imaging.

magnetic resonance imaging is considered the most noninvasive diagnostic method of detecting lesions of the intra-articular reliable knee structures. However, there are recent reports concluding that ultrasound is a valid technique for diagnosing meniscal lesions, even though it is not part of the standard protocol for evaluating injuries to the intra-articular knee structures.

DETAILED DESCRIPTION:
The aim of our study is to determine if any other available noninvasive method can reliably diagnose knee meniscal pathology as well as magnetic resonance imaging. In our case, we use ultrasound as a noninvasive method , and we want to see if this will be sufficient for diagnosing meniscal lesions , if it could be used for this task instead of magnetic resonance imaging investigations performed by a radiologist, as well as a guide for indication of knee arthroscopy .Knee ultrasound is widely accepted among orthopedic surgeons, and ultrasound is used as diagnostic tool for various pathological conditions in orthopedic surgery. ultrasound is currently popularly used in orthopedic surgery due to its simplicity and because it is less time-consuming and more practical than magnetic resonance imaging. It can diagnose location of the tear, joint effusion, synovial thickening, and osteophytosis. Rather, the goal is to determine whether or not meniscal pathology wanting surgical intervention .

We will also compare the diagnostic accuracies of these diagnostic procedures for both acute and chronic meniscal lesions of the knee.While magnetic resonance imaging (MRI) is often considered the gold standard diagnostic imaging modality for detection of meniscal abnormalities, it is associated with misdiagnosis in as high as 47% of cases, and is not readily available to a large number of patients. Ultrasonographic examination of the knee will be reported to be an effective diagnostic tool for this purpose with the potential to overcome many of the shortcomings of magnetic resonance imaging. The purpose of this study is to determine the clinical usefulness of ultrasonography for diagnosis of meniscal pathology in patients with acute knee pain and compare its diagnostic accuracy to magnetic resonance imaging in a clinical setting . Musculoskeletal ultrasound involves the use of high-frequency sound waves to image soft tissues and bony structures in the body for the purposes of diagnosing pathology . Recently, an increasing number of physicians have integrated musculoskeletal ultrasound into their practices to facilitate patient care. Technological advancements, improved portability, and reduced costs continue to drive the proliferation of ultrasound in clinical medicine the clinical applications of musculoskeletal ultrasound in clinical practice, including the ultrasonographic appearance of normal and abnormal tissues as well as specific diagnostic and interventional applications in major body regions.

ELIGIBILITY:
Inclusion Criteria:• Patients Presented with knee pain .

• High probability for requiring surgical intervention for diagnosis and/or treatment of the affected• Patients aged 14 years old and older. exclusion criteria. • Patients will be excluded when the criteria mentioned before not met. • When informed consent is not granted and documented .

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study willbe on cases of meniscal lesion degenerative on different pathologieslike osteoarthritis, rumatoid arthritis and trumatic cases due to meniscal injury these cases willbe diagnsed by ultrasound and compared by magnetic resonance imaging results to prove role of muskloskeletal ultrasound in diagnosis of meniscal lesions
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-05 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
rate of diagnosis of meniscal abnormalities | 48
  numbers of patient accurately diagnosed meniscal abnormality by ultrasound versus mri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Majewski M, Susanne H, Klaus S. Epidemiology of athletic knee injuries: A 10-year study. Knee. 2006 Jun;13(3):184-8. doi: 10.1016/j.knee.2006.01.005. Epub 2006 Apr 17. PMID 16603363
- [Background] Lee D, Bouffard JA. Ultrasound of the knee. Eur J Ultrasound. 2001 Oct;14(1):57-71. doi: 10.1016/s0929-8266(01)00146-x. No abstract available. PMID 11567855